CLINICAL TRIAL: NCT01434368
Title: A Longitudinal Investigation of the Endocrine and Neurobiologic Events Accompanying Puberty
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110251; 11-M-0251
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-09-25

CONDITIONS: fMRI
Keywords: Functional Magnetic Resonance Imaging (fMRI); Normal Development; Puberty; Natural History; Healthy Volunteer; HV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- children age 8-17 years admitted to pilot brain imaging studies: children age 8-17 years admitted to pilot brain imaging studies
- healthy adults: healthy adults ages 25 - 35 years at the time of enrollment
- typically developing children (with evidence of advanced bone age: typically developing children (with evidence of advanced bone age relative to chronologic age); age 8 or ages 12-13
- typically developing children ages 12/13 17 years: typically developing children ages 12 or 13 - 17 years
- typically developing children ages 8 17 years: typically developing children ages 8 - 17 years

SUMMARY:
Despite the clear importance of adolescence in the emergence of a number of disease states and processes, there is surprisingly little known about how the endocrine and metabolic events accompanying puberty in humans impact normal developmental neurobiology. Epidemiologic studies have identified sexual dimorphisms in the prevalence of several neuropsychiatric disorders, including depression, schizophrenia, and substance abuse. Many of these sex differences emerge during or shortly after puberty and are maintained until the 5th-6th decade of life. For example, the two-fold greater risk of unipolar depression in women compared with men does not appear until adolescence, and prior to puberty girls are not at increased risk relative to boys. Puberty is a structured, transitional process that can be influenced by both nutritional factors and environmental stressors; nonetheless, the variability in the timing and duration of puberty is largely determined by oligogenic inheritance. Basic neuroscience research has demonstrated that hormonal events accompanying puberty impact on many of the physiologic systems involved in the regulation of brain function (e.g., the appearance of new neurons in a brain-region specific pattern, neuronal remodeling, and the pruning of cortical connectivity). Additionally, not only does stress during puberty increase the risk of disturbances in affective adaptation during adulthood, but the events accompanying puberty modify stress responsivity (e.g., alterations in the duration and peak response of hypothalamic-pituitary-adrenal [HPA] axis hormones to stressors). Moreover, animal work has demonstrated that neural connectivity differs in a brain regional specific manner according to the stage of puberty (i.e., early versus late). In humans, puberty also occurs in stages, and although the endocrinology of puberty, surprisingly, has not been fully characterized with longitudinal data, studies have documented that the physical changes measured by Tanner stages I to V are accompanied by progressive increases in the secretions of both gonadal and adrenal steroids. Nonetheless, there remains considerable variability in the timing and duration of this otherwise highly structured reproductive transition.

We propose to perform a longitudinal, naturalistic study examining changes in brain structure and function, behavior, and stress responsivity in boys and girls across the pubertal transition. Because the pubertal transition is defined by a complex series of physiologic events that emerge sequentially over several years and involve changes in multiple endocrine and growth systems, and because there is also considerable variability in the timing of these events reflecting the influence of both genetic and environmental factors, puberty cannot by delineated by age of the participants as has been done in most imaging and other neurobiological studies of adolescence. The present study will formally bridge this gap by defining pubertal events per se in participants.

Participants will include healthy boys and girls whose pubertal status will be assessed, and in whom endocrine, metabolic, and brain imaging measures will be evaluated at eight - ten month intervals from age eight years (pre-puberty) until age 17 years (post-puberty). Reproductive endocrine, metabolic, and physical measures will be employed to characterize the stage and duration of pubertal development. Outcome measures will be derived via multimodal neuroimaging techniques, cognitive/behavioral assessments, metabolic measurements, and evaluations of HPA axis function. Additionally, the impact of genetic variation on the developmental trajectory of these parameters (both reproductive and CNS) will be determined.

This cross-institute proposal will employ a multidisciplinary approach to evaluating the effects on CNS function of the process of puberty in both boys and girls. This work will not only serve to inform research on the mechanisms by which sexual dimorphisms in neuropsychiatric disorders develop, it will also have important implications for the prevention and treatment of these disorders.

...

DETAILED DESCRIPTION:
Despite the clear importance of adolescence in the emergence of a number of disease states and processes, there is surprisingly little known about how the endocrine and metabolic events accompanying puberty in humans impact normal developmental neurobiology. Epidemiologic studies have identified sexual dimorphisms in the prevalence of several neuropsychiatric disorders, including depression, schizophrenia, and substance abuse. Many of these sex differences emerge during or shortly after puberty and are maintained until the 5th-6th decade of life. For example, the two-fold greater risk of unipolar depression in women compared with men does not appear until adolescence, and prior to puberty girls are not at increased risk relative to boys. Puberty is a structured, transitional process that can be influenced by both nutritional factors and environmental stressors; nonetheless, the variability in the timing and duration of puberty is largely determined by oligogenic inheritance. Basic neuroscience research has demonstrated that hormonal events accompanying puberty impact on many of the physiologic systems involved in the regulation of brain function (e.g., the appearance of new neurons in a brain-region specific pattern, neuronal remodeling, and the pruning of cortical connectivity). Additionally, not only does stress during puberty increase the risk of disturbances in affective adaptation during adulthood, but the events accompanying puberty modify stress responsivity (e.g., alterations in the duration and peak response of hypothalamic-pituitary-adrenal [HPA] axis hormones to stressors). Moreover, animal work has demonstrated that neural connectivity differs in a brain regional specific manner according to the stage of puberty (i.e., early versus late). In humans, puberty also occurs in stages, and although the endocrinology of puberty, surprisingly, has not been fully characterized with longitudinal data, studies have documented that the physical changes measured by Tanner stages I to V are accompanied by progressive increases in the secretions of both gonadal and adrenal steroids. Nonetheless, there remains considerable variability in the timing and duration of this otherwise highly structured reproductive transition.

We propose to perform a longitudinal, naturalistic study examining changes in brain structure and function, behavior, and stress responsivity in boys and girls across the pubertal transition. Because the pubertal transition is defined by a complex series of physiologic events that emerge sequentially over several years and involve changes in multiple endocrine and growth systems, and because there is also considerable variability in the timing of these events reflecting the influence of both genetic and environmental factors, puberty cannot by delineated by age of the participants as has been done in most imaging and other neurobiological studies of adolescence. The present study will formally bridge this gap by defining pubertal events per se in participants.

Participants will include healthy boys and girls whose pubertal status will be assessed, and in whom endocrine, metabolic, and brain imaging measures will be evaluated at eight - ten month intervals from age eight years (pre-puberty) until age 17 years (post-puberty). We will screen children in the clinic at age seven however will delay their first regular study visit until they are eight years old. Reproductive endocrine, metabolic, and physical measures will be employed to characterize the stage and duration of pubertal development. Outcome measures will be derived via multimodal neuroimaging techniques, cognitive/behavioral assessments, metabolic measurements, and evaluations of HPA axis function. Additionally, the impact of genetic variation on the developmental trajectory of these parameters (both reproductive and CNS) will be determined. These child participants will be offered the opportunity to return as adults. The data obtained from this unique sample will serve as an important self-as-own comparison of adult neuroimaging data in comparison to those data obtained across the pubertal transition (i.e., during adolescence). This will serve to extend the longitudinal data to include an adult end point.

This cross-institute proposal will employ a multidisciplinary approach to evaluating the effects on CNS function of the process of puberty in both boys and girls. This work will not only serve to inform research on the mechanisms by which sexual dimorphisms in neuropsychiatric disorders develop, it will also have important implications for the prevention and treatment of these disorders.

ELIGIBILITY:
* INCLUSION CRITERIA - SAMPLE 1:

Child volunteers will qualify for inclusion if they meet the following criteria:

* Good general health and normal IQ; A normal IQ will be determined by the scores on Test of Irregular Word Reading Efficiency (TIWRE)
* Age 8 years;
* Body Mass Index (kg/m^2) between the 15th and 85th percentiles for age and sex according to the US Centers for Disease Control and Prevention 2000 growth charts;
* A normal tempo of growth as determined by skeletal age within +/- 1.64 standard deviations of chronologic age according to the Greulich and Pyle radiographic atlas (i.e., no evidence for precocious puberty or abnormal delay of maturation); Research criteria for determining bone age will be performed by the collaborating pediatric endocrinologist. This criterion is required only for the initial entry into this study and is not one of the inclusion criteria for subsequent visits;
* No history of significant neurologic or cognitive disorders. Examples include neonatal anoxic encephalopathy, seizure disorders, autism, and most learning disorders including attention deficit hyperactivity disorder;
* Able to provide assent. Parents will provide consent.
* Able to speak and read English.

EXCLUSION CRITERIA - SAMPLE 1:

Child volunteers will be excluded for the following reasons:

* Presence of any medical condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in eye or other body part, dental braces);
* Presence or history of medical conditions known to affect cerebral anatomy;
* Children who are not pre-pubertal as indicated by the presence of Tanner stage 2 development (i.e., areolar development in girls and testicular volume > 3 cc in boys);
* Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or any other condition which, in the opinion of the investigators, would impede the ability to give informed consent or possibly hinder completion of the study; presence of any psychiatric disorder in the subject, sibling, or other first-degree relative;
* Subjects who regularly use prescription medications (the use of over-the-counter medications will be reviewed on a case-by-case basis.);
* For females who have reached menarche: Pregnancy, lactation, or inability or unwillingness to undergo pregnancy testing (a urine pregnancy test will be performed prior to all MRI and X-ray procedures for girls who have had the onset of menses);
* Current or past use of psychiatric medication;
* I.Q. < 70 (determined by the scores on Test of Irregular Word Reading Efficiency [TIWRE]).

INCLUSION CRITERIA - SAMPLE 2:

Child volunteers will qualify for inclusion if they meet the following criteria:

* Good general health and normal IQ; A normal IQ will be determined by the scores on Test of Irregular Word Reading Efficiency (TIWRE)
* Ages 12-13 years;
* Body Mass Index (kg/m^2) between the 15th and 85th percentiles for age and sex according to the US Centers for Disease Control and Prevention 2000 growth charts;
* A normal tempo of growth as determined by skeletal age within +/- 1.64 standard deviations of chronologic age according to the Greulich and Pyle radiographic atlas (i.e., no evidence for precocious puberty or abnormal delay of maturation); Research criteria for determining bone age will be performed by the collaborating pediatric endocrinologist. This criterion is required only for the initial entry into this study and is not one of the inclusion criteria for subsequent visits.;
* No history of significant neurologic or cognitive disorders. Examples include neonatal anoxic encephalopathy, seizure disorders, autism, and most learning disorders including attention deficit hyperactivity disorder;
* Able to provide assent. Parents will provide consent.
* Able to speak and read English.

EXCLUSION CRITERIA - SAMPLE 2:

Child volunteers will be excluded for the following reasons:

* Presence of any medical condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in eye or other body part, dental braces);
* Presence or history of medical conditions known to affect cerebral anatomy;
* Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or any other condition which, in the opinion of the investigators, would impede the ability to give informed consent or possibly hinder completion of the study; presence of any psychiatric disorder in the subject, sibling, or other first-degree relative;
* Subjects who regularly use prescription medications (the use of over-the-counter medications will be reviewed on a case-by-case basis.);
* For females who have reached menarche: Pregnancy, lactation, or inability or unwillingness to undergo pregnancy testing (a urine pregnancy test will be performed prior to all MRI and X-ray procedures for girls who have had the onset of menses);
* Current or past use of psychiatric medication;
* I.Q. < 70 (determined by the scores on Test of Irregular Word Reading Efficiency [TIWRE]).

INCLUSION/EXCLUSION CRITERIA - SAMPLE 3:

Inclusion and exclusion criteria for sample 3 will be identical as those for sample 2 with the exception that children between the ages of 8 and 17 will be included.

INCLUSION/EXCLUSION CRITERIA - SAMPLE 4:

Sample 4 participants will also be volunteering in Protocol #95-M-0150 Neurobiological Investigation of Patients with Schizophrenia Spectrum Disorders and Their Siblings, and/or Protocol #81-M-0126, The Evaluation of Women with Menstrually-Regulated Mood and Behavioral Disorders, in which they will also have signed consent and through which they will have been screened.

INCLUSION CRITERIA - SAMPLE 4:

* Ages of 25 to 35 years at the time of enrollment.
* Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
* No use of psychotropic substances in the last 3 months.
* No psychiatric or severe chronic medical illness at the time of the study, and by history.
* Able to speak and read English.

EXCLUSION CRITERIA - SAMPLE 4:

* Presence of impaired hearing.
* Pregnant or currently breast feeding. (a urine pregnancy test will be performed prior to MRI procedures in women).
* Presence of a history head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma.
* Previous eye surgery with a prosthetic implant.
* Participants with tattoos will be excluded if the tattoos are in a location on the body (eyes, lips, etc.) that could interfere with fMRI scans or contain a heavy metal content.
* Presence of any non-organic implant or any other device such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitro), any metallic implants or objects, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunt.
* Presence of cerebral or other aneurysm clips.
* Presence of shrapnel or other metal imbedded in the body (such as from war wounds or accidents).
* Previous employment in metal fields or with machines that may have left any metallic fragments in or near the eyes.
* History of a severe accident in the past that may possibly have left metal in the body.
* Psychological contraindications for MRI (e.g., suffer from claustrophobia);
* Less than an 8th grade education or an IQ below 70 as determined by the scores on Test of Irregular Word Reading Efficiency [TIWRE] .

INCLUSION/EXCLUSION CRITERIA - SAMPLE 5:

Inclusion and exclusion criteria for sample 5 will be identical as those for samples 1 and 2 (i.e., children will either be age 8-9 or between the ages of 12 and 13) with the exception that children with a tempo of growth that is considered abnormal as demonstrated by skeletal age greater than two standard deviations in advance of their chronologic age according to the Greulich and Pyle Radiographic Atlas will be included. These children will be matched for age, Tanner stage, race, ethnicity, and BMI with children currently enrolled in the longitudinal study.

SAMPLE 6

Participants will have participated in this protocol as children in either Sample 1 or sample 2.

INCLUSION CRITERIA:

* Age 19 to 30 years at the time of re-enrollment.
* Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
* Normal physical exam, routine labs and absence of axis 1 psychiatric illnesses as confirmed by a Structured Diagnostic Interview for DSM-5 (SCID).
* No current use of psychotropic substances.

EXCLUSION CRITERIA:

* Presence of any implant or medical condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in eye or other body part, dental braces);
* Presence or history of medical conditions known to affect cerebral anatomy;
* Individuals who have current substance abuse or a psychiatric disorder or any other condition which, in the opinion of the investigators, would impede the ability to give informed consent or possibly hinder completion of the study;
* Current use of psychiatric medication or presence of any psychiatric disorder;
* For females: pregnancy, lactation, or inability or unwillingness to undergo pregnancy testing (a urine pregnancy test will be performed prior to all MRI procedures);

Ages: 7 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Total requested accrual Total expected accrual for all groups: 370 This total is comprised of the following groups: 280 typically developing children ages 8 17 years, boys (n = 140); girls (n = 140) 20 typically developing children (with evidence of advanced bone age relative to chronologic age); age 8 or ages 12-13 50 healthy adults ages 25 35 years at the time of enrollment, men (n = 25); women (n = 25) 20 children age 8-17 years admitted to pilot brain imaging studies
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2011-11-23 (Actual)

PRIMARY OUTCOMES:
fMRI BOLD signal | ongoing
  fMRI BOLD signal

SECONDARY OUTCOMES:
structural MRI findings, DTI, UFC, | ongoing
  structural MRI findings, DTI, UFC

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Ogunleye OA, Raviprakash H, Simmons AM, Bovell RTM, Martinez PE, Yanovski JA, Berman KF, Schmidt PJ, Jones EC, Bagheri H, Biassou NM, Hsu LY. A Combined Region- and Pixel-Based Deep Learning Approach for Quantifying Abdominal Adipose Tissue in Adolescents Using Dixon Magnetic Resonance Imaging. Tomography. 2023 Jan 15;9(1):139-149. doi: 10.3390/tomography9010012. PMID 36648999
- [Derived] Cole KM, Wei SM, Martinez PE, Nguyen TV, Gregory MD, Kippenhan JS, Kohn PD, Soldin SJ, Nieman LK, Yanovski JA, Schmidt PJ, Berman KF. The NIMH Intramural Longitudinal Study of the Endocrine and Neurobiological Events Accompanying Puberty: Protocol and rationale for methods and measures. Neuroimage. 2021 Jul 1;234:117970. doi: 10.1016/j.neuroimage.2021.117970. Epub 2021 Mar 24. PMID 33771694
- [Derived] Chen G, Nash TA, Cole KM, Kohn PD, Wei SM, Gregory MD, Eisenberg DP, Cox RW, Berman KF, Shane Kippenhan J. Beyond linearity in neuroimaging: Capturing nonlinear relationships with application to longitudinal studies. Neuroimage. 2021 Jun;233:117891. doi: 10.1016/j.neuroimage.2021.117891. Epub 2021 Mar 3. PMID 33667672
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-M-0251.html